CLINICAL TRIAL: NCT01676480
Title: The Effect of Endurance Training on Body Composition and Insulin Sensitivity in Prostate Cancer Patients Receiving ADT
Brief Title: The Effect of Endurance Training on Body Composition and Insulin Sensitivity in Prostate Cancer Patients Receiving Androgen Deprivation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inge Holm (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Sponsor-Investigator, Inge Holm, Administrator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-4-2009-102
Record Dates: First submitted 2012-01-10; First posted 2012-08-31 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; ADT; Endurance training
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Endurance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ADT group (Experimental)
  Interventions: Behavioral: Endurance training
- Control group (Experimental)
  Interventions: Behavioral: Endurance training

INTERVENTIONS:
Behavioral: Endurance training — 12 weeks of endurance training 3 times per week

SUMMARY:
The purpose of the present study is to investigate if endurance training can be used as a therapeutic action against the adverse metabolic disturbances and unfavourable changes in body composition that accompany the androgen deprivation therapy (ADT) treatment in prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients receiving ADT for at least 3 months
* Healthy age and BMI matched controls

Exclusion Criteria:

* severe cardiovascular disease
* severe arthritis
* severe neuropathy
* severe hypertension
* therapy with antidiabetic agents
* VO2max > 30.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Changes in body composition and insulin sensitivity in response to training | Body composition and insulin sensitivity are measured at baseline and after 12 weeks of endurance training

CONTACTS AND LOCATIONS:
Overall Officials: Bente K Pedersen, Study Director — Centre of Inflammation and Metabolism, Rigshospitalet
Locations (1):
- Centre of Inflammation and Metabolism, Rigshospitalet, Copenhagen, Denmark